CLINICAL TRIAL: NCT07125027
Title: A Multicomponent Intervention for Patients With Lumbosacral Radiculopathy: Move-MORE
Acronym: Move-MORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Oregon Health and Science University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Ryan Wexler, Assistant Research Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RW6625; K12NS130673 (NIH)
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Lumbosacral Radiculopathy; Sciatica; Chronic Low Back Pain With a Neuropathic Component; Radiculopathy Lumbar; Chronic Pain (Back / Neck)
Keywords: Mindfulness; Physical Activity; Motivational Interviewing; Meditation; Tai Chi/Qi Gong; Movement; Mindfulness-Oriented Recovery Enhancement; Mindfulness-Based Interventions; Radiculopathy; Lumbosacral Radiculopathy; Lumbar Radiculopathy; Chronic low back pain; Low back pain; Back Pain
MeSH Terms: conditions — Sciatica; Chronic Pain; Motor Activity; Radiculopathy; Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will go through the multicomponent Move-MORE program. Move-MORE is an integrated mind-body intervention which combines mindfulness, physical activity, and motivational interviewing informed by the principles of self-determination theory
  Interventions: Behavioral: Move-MORE

INTERVENTIONS:
Behavioral: Move-MORE — Move-MORE is a multicomponent intervention which combines mindfulness training, physical activity, and motivational interviewing informed by the principles of self-determination theory. The version of Move-MORE being used in this study is specifically designed for use in patients with lumbosacral radiculopathy.

SUMMARY:
The Move-MORE study is designed to evaluate a multicomponent mindfulness and movement program for patients with lumbosacral radiculopathy. The program brings together mindfulness training to help participants develop awareness of their body and manage pain-related stress, gentle movement practice to improve comfort with physical activity and support function, and motivational interviewing to strengthen motivation, confidence, and the ability to make healthy changes.

The main objectives are to determine whether it is feasible for participants to use each component of the program when delivered online, to assess how acceptable and engaging each component is, and to evaluate the impact on pain, physical function, and daily activity levels. The study intervention will be conducted entirely remotely. Participants will complete online surveys, brief daily check-ins on their phone, and wear a small activity monitor on the hip to measure movement. They will also undergo quantitative sensory testing to evaluate pain sensitivity. At the end of the program, participants will share feedback about their experiences via qualitative interviews.

The findings will help identify which parts of the program provide the greatest benefit, with the ultimate goal of developing a more targeted and effective digital program for people with this condition.

DETAILED DESCRIPTION:
Lumbosacral radiculopathy (LR) is a spinal pathology that manifests as pain, weakness, and numbness in the lower extremity. Commonly referred to as "sciatica", LR has a lifetime prevalence up to 43%, and can often become an intractable condition with long-term outcomes unimproved by conventional biomedical treatments such as surgery. Thus, we seek to develop a non-invasive and non-pharmacologic treatment for LR patients

This study aims to 1) develop a multicomponent intervention that integrates Mindfulness-Oriented Recovery Enhancement and physical activity for patients with LR, 2) assess the feasibility and acceptability of this multicomponent intervention, and 3) evaluate preliminary efficacy of the intervention via self-report measures of pain, disability, kinesiophobia, and other psychosocial factors related to chronic pain. In addition, this study will use quantitative sensory testing (i.e., pressure and heat pain thresholds) as an objective measure of pain.

The multicomponent intervention will be developed (AIM 1) using qualitative data from focus groups of LR patients and semi-structured interviews from a multidisciplinary sample of physicians who treat LR. This data will be analyzed using a thematic approach to assess barriers and facilitators to participation, patients' perspectives on non-pharmacologic interventions, and physicians' views of medically necessary considerations. Qualitative findings will be presented to a team of expert mindfulness instructors to support program design. In a single arm trial designed to assess feasibility, acceptability, and preliminary efficacy of the intervention (AIMS 2 and 3), we will administer the multicomponent program developed in Aim 1. Data will be collected from participants at three time points: baseline, midpoint, post-intervention, 3-month follow-up. In addition, ratings of pain intensity will be captured daily via ecologic momentary assessment.

During the intervention period, participants will be asked to attend virtual classes once a week. Between weekly sessions, participants will also be asked to track their home practice, daily levels of pain, and any adverse events via a daily survey. At the end of the study, participants will be asked to participate in a semi-structured exit interview which will inquire about their experience in the intervention.

This study seeks to shift the current research paradigm by being the first to develop and test a novel non-invasive, non-pharmacologic, multicomponent intervention for LR. As such, the proposed research contributes much needed scientific knowledge toward identifying efficacious treatments for a highly prevalent, costly, and intractable condition.

ELIGIBILITY:
Inclusion Criteria:

* ● Adults age 18-65 years at the time of enrollment

  * Ability to stand for 10 minutes
  * Presence of lumbosacral radicular pain within the past week that extends below the knee (i.e., pain radiating from the low back into the leg in a nerve root distribution) with or without accompanying low back pain, of at least 12 weeks' duration, AND
  * Tampa Scale of Kinesiophobia score ≥ 23
  * At least one positive physical examination finding consistent with lumbosacral radiculopathy, including at least one of the following:

    * Positive straight leg raise test (eliciting radicular pain below the knee at ≤70 degrees of elevation);
    * Positive Valsalva maneuver (eliciting radiculcar pain below the knee);
    * Positive slump test;
    * Neurological deficit in a lumbar nerve root distribution, including at least one of the following:

      * Dermatomal sensory loss,
      * Myotomal weakness, or
      * Reduced or absent deep tendon reflexes (e.g., patellar or Achilles reflex) corresponding to the affected nerve root.
  * Daily access to the internet via cell phone, tablet, or computer
  * Willing to engage with Move-MORE 4-5 times per week on your own
  * Willing to attend a two-hour-long virtual Zoom meeting once per week for eight weeks
  * Willing to attend two in-person study visits and a follow-up visit
  * Willing to complete 18 questionnaires pertaining to your pain symptoms, quality of life, psychosocial experiences, and your experiences in the trial
  * Willing to wear an actigraphy device all day, every day, and while sleeping, for the duration of study participation and willing to keep it charged
  * Willing to respond to a daily online survey for the duration of study participation
  * Able to speak, read, and understand the English language
  * Able to provide written informed consent
  * Moderately motivated to participate as reported on a numeric rating scale (≥ 4/10)

Exclusion Criteria:

* ● Participants will be excluded if they have clinical signs or symptoms of lumbosacral radiculopathy with progressive neurologic deficits (loss of motor or sensory function) or intolerable pain.

  * Participants with lumbosacral radiculopathy with progressive neurologic deficits will be referred for immediate medical attention, and are not eligible for participation in this study.

    ● Participants will be excluded if they have clinical signs or symptoms suggestive of cauda equina syndrome, including any of the following:
  * New-onset urinary retention or overflow incontinence not attributable to other known causes;
  * Fecal incontinence;
  * New onset of saddle anesthesia (loss of sensation in the buttocks, perineum, and inner thighs);
  * Severe or progressive bilateral lower extremity weakness;

    * Participants with suspected cauda equina syndrome will be referred for immediate medical attention, and are not eligible for participation in this study.

      * Presence of moderate to severe foot drop, defined as noticeable weakness in ankle dorsiflexion that interferes with walking or requires the use of an assistive device (e.g., ankle-foot orthosis). Participants with suspected or worsening foot drop will be referred for further evaluation and are not eligible for study participation.
      * Current use of a spinal cord stimulator
      * Have received epidural steroid injection in the prior 3 months
      * Have received a surgical intervention for low back pain or lumbosacral radiculopathy in the previous 6 months
      * Current active mindfulness meditation practice 1 time/week or more, and/or history of formal training in mindfulness/meditation practice
      * Concurrent diagnosis of cancer
      * Current unmanaged or uncontrolled mental illness known to cause psychosis: schizophrenia, schizotypal disorders, bipolar I disorder with psychosis, major depressive disorder with psychosis
      * Diagnosis of Borderline Personality Disorder or score >6 on the McLean Screening Instrument for Borderline Personality Disorder
      * Initiation of or changes to an exercise regimen within 2 weeks prior to screening and/or enrollment
      * Major medical or surgical event requiring hospitalization (for any reason other than a minor scheduled medical procedure) within 3 months prior to screening; or, scheduled or will be scheduled to occur within the 20 weeks (i.e., five months) after enrollment
      * Currently participating in another interventional research study or participated in another interventional study within 2 weeks prior to screening
      * Any reason the Clinical Investigator or Principal Investigator believes confers increased risk to the potential participant, if they were to enroll in the study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | Week 0, Week 4, Week 8, Week 20
  Activities of daily living. Min = 0%, Max = 100%. Higher score = worse outcomes.

SECONDARY OUTCOMES:
painDETECT Questionnaire | Week 0, Week 4, Week 8, Week 20
  Neuropathic Pain. Min = -1, Max = 38. Higher score = worse outcomes.
Client Satisfaction Questionnaire | Week 4, Week 8, Week 20
  Intervention Satisfaction. Min = 8, Max = 32. Higher score = greater satisfaction.
Visual Analog Scale | Daily
  Pain Intensity. Min = 0, Max = 10. Higher score = worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author, R.S.W., upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2027-
Access Criteria: The data that support the findings of this study are available from the corresponding author, R.S.W., upon reasonable request.

REFERENCES:
- See also: Helfgott Research Institute - Join a Study — https://nunm.edu/research/study-opportunities/
- See also: Helfgott Research Institute - Projects — https://nunm.edu/research/projects/